CLINICAL TRIAL: NCT07192471
Title: A Phase 1, Multicenter, Open-label, Non-randomized, Dose-escalation and Backfill Study of KK2223 in Participants With Relapsed or Refractory T-cell Non Hodgkin Lymphoma
Brief Title: A First-in-Human Study of KK2223 in Participants With Relapsed or Refractory T Cell Non-Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2223-001
Record Dates: First submitted 2025-08-12; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: T-cell NHL (PTCL or CTCL)
Keywords: Neoplasms; Lymphoma; Immune System Diseases; First in Human; Lymphoma, T-Cell, Cutaneous +; Lymphoma, T-Cell, Peripheral; Mycosis fungoides; Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Neoplasms; Lymphoma; Immune System Diseases; Lymphoma, T-Cell, Peripheral; Mycosis Fungoides; Sezary Syndrome

STUDY DESIGN:
Intervention Model Description: This is a sequential design study where participants receive interventions in a stepwise manner. Treatment assignments and doses may be adjusted based on interim safety and efficacy analyses conducted throughout the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part One (Dose Escalation) (Experimental): In Part 1, safety and tolerability of KK2223 in relapsed/refractory PTCL or CTCL patients will be assessed using a BOIN dose-escalation design.
  Interventions: Drug: KK2223
- Part Two (Backfill) (Experimental): Part 2 will collect additional data, with dose levels and cohort size based on Part 1 results, administering doses approved for tolerability. Backfill cohorts at cleared doses may open, prioritizing Part 1 enrollment.
  Interventions: Drug: KK2223

INTERVENTIONS:
Drug: KK2223 — Intravenous infusion

SUMMARY:
The purpose of this study is to determine the safety, tolerability, PK and pharmacodynamics of KK2223 in adult participants with relapsed or refractory peripheral T cell lymphoma (PTCL) or cutaneous T cell lymphoma (CTCL).

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label, non randomized study in participants with relapsed or refractory PTCL or CTCL. This study consists of Part 1 (dose-escalation) and Part 2 (backfill). The purpose of this study is to determine the safety, tolerability, PK and pharmacodynamics of K2223 in r/r T-cell NHL (PTCL or CTCL)

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with confirmed T-cell lymphoma subtypes: PTCL (including nodal T-follicular helper cell lymphoma, ALCL, PTCL NOS) for Parts 1 and 2; CTCL (mycosis fungoides and Sézary syndrome, stages IIB-IV) for Parts 1 and 2, with specific disease involvement criteria in Part 2.
* PTCL participants must have relapsed/refractory/intolerant to ≥1 systemic therapy; CD30+ PTCL must have prior brentuximab vedotin treatment or intolerance, and/or ALK-positive ALCL participants should have previously received crizotinib if indicated (crizotinib administration is applicable to US sites only). CTCL participants must have relapsed/refractory/intolerant to ≥2 systemic therapies.
* Availability of tumor tissue (current or archival) is required.
* Measurable disease required: nodal/extranodal lesions for PTCL and assessable skin disease for CTCL.
* ECOG performance status 0-1; adequate neutrophils (≥1000/µL), platelets (≥75,000/µL), renal function (creatinine clearance ≥60 mL/min), liver function within defined limits, and total bilirubin ≤1.5× ULN (up to 3× ULN with Gilbert's syndrome).
* Life expectancy ≥3 months.
* Negative pregnancy test for females of childbearing potential; contraception required for females and males with partners of childbearing potential during and after treatment.
* Restrictions on gamete donation and freezing during and after treatment.
* Ability to provide informed consent and comply with study procedures. -

Exclusion Criteria:

* Recent autologous or allogeneic transplant within 120 days before treatment; active GVHD or ongoing immunosuppression after allogeneic transplant.
* Pregnant or breastfeeding females, or those intending pregnancy; males with partners intending pregnancy.
* History of HIV, HBV, or HCV infections generally excluded, except for controlled or resolved cases as defined.
* Uncontrolled infections requiring IV antibiotics, antivirals, or antifungals at screening through treatment start.
* Significant medical history or complications within six months prior to enrollment, including advanced congestive heart failure (NYHA Class III or higher), recent unstable angina or myocardial infarction, autoimmune diseases requiring systemic immunosuppressive therapy, active or uncontrolled ocular diseases, Grade 3 or 4 peripheral neuropathy, or other poorly controlled conditions as judged by the investigator (e.g., uncontrolled hypertension, diabetes, or arrhythmias).
* Use of other investigational drugs within 14 days or 5 half-lives before treatment.
* Steroid use over 10 mg/day prednisone equivalent within 14 days prior, except limited corticosteroid use with specific tapering guidelines; topical steroids allowed under conditions for CTCL.
* Major surgery, radiotherapy, chemotherapy, or other anti-cancer treatments within 14 days or 5 half-lives before treatment.
* Prior mogamulizumab use within six months before treatment; associated rash must be ruled out if >6 months.
* Failure to recover from prior non-hematologic toxicities to Grade 0 or 1 (except alopecia and mild neuropathy).
* Prolonged QT/QTc interval (e.g., QTcF >480 ms).
* Active second primary malignancies except specified non-exclusionary cases.
* CNS involvement.
* Any condition that may impair compliance or study completion as judged by the Investigator.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Assess the incidence of treatment-emergent adverse events and determine the maximum tolerated dose (MTD) of KK2223 in patients with relapsed or refractory peripheral or cutaneous T cell lymphoma (PTCL/CTCL). | Through study completion, an average of 1.5 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 (all 72 potentially treated subjects)
Assess the incidence of treatment-emergent adverse events and determine the maximum tolerated dose (MTD) of KK2223 in patients with relapsed or refractory peripheral or cutaneous T cell lymphoma (PTCL/CTCL). | Through study completion, an average of 1.5 years
  Vital signs (mmHg in Systolic/Diastolic blood pressure)
Assess the incidence of treatment-emergent adverse events and determine the maximum tolerated dose (MTD) of KK2223 in patients with relapsed or refractory peripheral or cutaneous T cell lymphoma (PTCL/CTCL). | Through study completion, an average of 1.5 years
  Pulse rate (beats/min)
Assess the incidence of treatment-emergent adverse events and determine the maximum tolerated dose (MTD) of KK2223 in patients with relapsed or refractory peripheral or cutaneous T cell lymphoma (PTCL/CTCL). | Through study completion, an average of 1.5 years
  Respiratory Rate (breath/min)
Assess the incidence of treatment-emergent adverse events and determine the maximum tolerated dose (MTD) of KK2223 in patients with relapsed or refractory peripheral or cutaneous T cell lymphoma (PTCL/CTCL). | Through study completion, an average of 1.5 years
  Temperature (°Celcius)
Assess the incidence of treatment-emergent adverse events and determine the maximum tolerated dose (MTD) of KK2223 in patients with relapsed or refractory peripheral or cutaneous T cell lymphoma (PTCL/CTCL). | Through study completion, an average of 1.5 years
  ECG parameters (PR interval, QRS interval, QT interval, QTc interval)
Assess the incidence of treatment-emergent adverse events and determine the maximum tolerated dose (MTD) of KK2223 in patients with relapsed or refractory peripheral or cutaneous T cell lymphoma (PTCL/CTCL). | Through study completion, an average of 1.5 years
  Number of participants with dose-limiting toxicities (DLTs) in Part 1 only (at most 27 participants) and assess maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
To evaluate the blood drug concentration | Through study completion, an average of 1.5 years
To evaluate the immunogenicity of KK2223. | Through study completion, an average of 1.5 years
  Incidence of Anti drug antibodies (ADA) in blood
To evaluate the preliminary anti-tumor activity of KK2223 (Investigator assessed). | Through study completion, an average of 1.5 years
  % in Overall Response Rate (ORR)
To evaluate the preliminary anti-tumor activity of KK2223 (Investigator assessed). | Through study completion, an average of 1.5 years
  % in Compartment Response (if applicable)
To evaluate the preliminary anti-tumor activity of KK2223 (Investigator assessed). | Through study completion, an average of 1.5 years
  Time unit (week/month) in Duration of Response (DOR)
To evaluate the preliminary anti-tumor activity of KK2223 (Investigator assessed). | Through study completion, an average of 1.5 years
  Time unit (week/month) in Time To Next Treatment (TTNT) will be evaluated
To evaluate the preliminary anti-tumor activity of KK2223 (Investigator assessed). | Through study completion, an average of 1.5 years
  Time unit (week/month) in Time To Response (TTR)

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the study sponsored by Kyowa Kirin will be available in the Vivli repository, https://vivli.org/ourmember/kyowa-kirin/ as long as conditions of data disclosure specified in the policy section of the Vivli website are satisfied.